CLINICAL TRIAL: NCT04205305
Title: Outcome in Patients Treated with Intraarterial Thrombectomy - OptiMAL Blood Pressure Control (OPTIMAL-BP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2019-1208
Record Dates: First submitted 2019-11-21; First posted 2019-12-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke
Keywords: Acute ischemic stroke; blood pressure; hypertension; endovascular thrombectomy; recanalization
MeSH Terms: conditions — Ischemic Stroke; Hypertension | interventions — Labetalol; Nicardipine

STUDY DESIGN:
Intervention Model Description: 1. The study is a multicenter, prospective, randomized, open-label trial with blinded end-point assessment (PROBE) design study.
  2. After successful revascularization, the active blood pressure control group and the standard blood pressure control group will be randomized by 1: 1.
  3. Patients who have undergone intraarterial thrombectomy due to acute cerebral infarction and have successfully reopened arteries will be enrolled.
  4. Medical history, laboratory findings and blood pressure parameters (systolic blood pressure, diastolic blood pressure, blood pressure variability, etc.), neurological scores, functional recovery, and quality of life indicators will be collected.
  5. Neurological scores, functional recovery scores, and quality of life indicators are performed by independent researchers in the blind state.
  6. All data is collected using e-CRF, and the image study will be anonymized and sent to the central adjudication.
Who Masked: Outcomes Assessor
Masking Description: Three months after discharge, the independence assessment will be performed by the researcher who don't know the patients group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional blood pressure control group (Active Comparator): systolic blood pressure <180 mmHg
  Interventions: Drug: conventional blood pressure control (labetalol, nicardipine)
- Intensive blood pressure control group (Experimental): systolic blood pressure <140 mmHg
  Interventions: Drug: intensive blood pressure control (labetalol, nicardipine)

INTERVENTIONS:
Drug: conventional blood pressure control (labetalol, nicardipine) — After successful recanalization, appropriate antihypertension medication is administered to control systolic blood pressure <180 mmHg.
  Arms: Conventional blood pressure control group
Drug: intensive blood pressure control (labetalol, nicardipine) — After successful recanalization, appropriate antihypertension medication is administered to control systolic blood pressure <140 mmHg.
  Arms: Intensive blood pressure control group

SUMMARY:
Recent endovascular thrombectomy (EVT) trial have proven the effectiveness of intraarterial revascularization in patients with larger cerebral artery occlusion. The success rate of EVT is close to 80%, but only 50% of patients improve to independent functional outcome. Therefore, new treatment strategies are needed to reduce the futile revascularization. However, updated guidelines recommend the indications for EVT based on the results of randomized clinical trials (RCT), management of post-revascularization is largely unknown.

Current guidelines suggest that systolic blood pressure should be adjusted below 180 mmHg and diastolic blood pressure below 105 mmHg in patients undergoing intraarterial reopening. However, in the case of successful recanalization by EVT, same guideline is adopted even though the possibility of intracerebral hemorrhage or reperfusion injury by high blood pressure. On the other hand, too low blood pressure can worsen cerebral ischemia.

Therefore, this study will compare the effectiveness of active blood pressure control group (with less than 140 mmHg systolic blood pressure) versus standard blood pressure control group (with less than 180 mmHg systolic blood pressure) during the first 24 hours in patients who underwent EVT and achieved successful recanalization (TICI 2b-3). The goal is to reach the target blood pressure within 60 minutes of randomization.

DETAILED DESCRIPTION:
1. The study is a multicenter, prospective, randomized, open-label trial with blinded end-point assessment (PROBE) design study.
2. After successful revascularization, the active blood pressure control group and the standard blood pressure control group will be randomized by 1: 1.
3. Patients who is admitted to the Department of Neurology at the participating hospital with acute cerebral infarction will will be included for 5 years from December 2019 to December 2023 (based on the date of stroke). Patients who have undergone intraarterial thrombectomy and have successfully reopened arteries should be enrolled.
4. Collect medical history, laboratory findings and blood pressure parameters (systolic blood pressure, diastolic blood pressure, blood pressure variability, etc.), neurological scores, functional recovery, and quality of life indicators.
5. Neurological scores, functional recovery scores, and quality of life indicators are performed by independent researchers in the blind state.
6. All data is collected using e-CRF, and the image study will be anonymized and sent to the central adjudication.
7. Central adjudication will review the image study.
8. One intermediate analysis will be conducted at the end of first period or when a half of study patients were enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20 years
2. Acute ischemic stroke patients who underwent intraarterial treatment for large vessel occlusion. (ICA, MCA M1 or M2, ACA A1, PCA P1)
3. Patients with successful recanalization after intraarterial thrombectomy (TICI 2b or TICI 3) 4. Patients with elevated BP (systolic BP ≥140 mmHg) on at least two measurements with a two-minute interval within 2 hours of successful recanalization.

Exclusion Criteria:

1. Age <20
2. Patients with contraindication for use antihypertensive medication after intraarterial thrombectomy.
3. Patients with blood pressure <140 mmHg after successful recanalization.
4. Patients with symptomatic intracranial hemorrhage after successful recanalization
5. Patients with pre-morbid neurological dysfunction (modified Rankin Scale, mRS >2)
6. Patients with severe medical and surgical diseases.
7. Patients who are considered having a difficulty to enrollment.
8. No informed consents from patients.
9. Patients who participated in a study that did not allow duplicate participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-07-23 (Actual); Study Completion 2023-07-23 (Actual)

PRIMARY OUTCOMES:
Modified Rankin scale scores(mRS) | 90 days
  Effectiveness outcome: Functional independence (modified Rankin score 0 to 2)
  -The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.
symptomatic intracerebral hemorrhage: Number of participants with symptomatic intracerebral hemorrhage | 36 hours
  Safety outcome: The definition in the European Cooperative Acute Stroke Study III (ECASS 3) will be adopted : a large local or remote parenchymal pattern (>30% of the infarcted area affected by hemorrhage, with mass effect or extension outside the infarct), intraventricular hemorrhage, or subarachnoid hemorrhage which is identified as the predominant cause of the neurologic deterioration from baseline (increase of ≥4 points in the NIHSS score) or death within 36 hours.
Death related to the index stroke within 90 days | 90 days

SECONDARY OUTCOMES:
BP parameters - systolic blood pressure | 24 hour
  change in systolic blood pressure
BP parameters - diastolic blood pressure | 24 hour
  change in diastolic blood pressure
BP parameters - blood pressure variability | 24 hour
  change in blood pressure variability
Functional independence | 1 month
  modified Rankin score 0 to 2
Distribution of the modified Rankin scores (shift analysis) | 90 days
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.
National Institutes of Health Stroke Scale(NIHSS) score | 24 hour
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.
Excellent recovery | 24 hour
  NIHSS 0 -1 or improvement more than 8. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.
Recanalization status on CT Angiography(CTA) or MR Angiography(MRA) | 24±12 hour
  occurence of TICI 2b or 3 recanalization on CTA or MRA
  - The thrombolysis in cerebral infarction(TICI) scale is a tool for determining the response of thrombolytic therapy for ischemic stroke. The original description 1 was based on the angiographic appearances of the treated occluded vessel and the distal branches(Grade 0: no perfusion, Grade 1: penetration with minimal perfusion, Grade 2: partial perfusion, Grade 2A: only partial filling(less than two-thirds) of the entire vascular territory is visualized, Grade 2B: complete filling of all of the expected vascular territory is visualized but the filling is slower than normal, Grade 3: complete perfusion)
Quality of life measured by Euro-QoL | 90 days
  EuroQol-5D (EQ-5D) is an instrument for measuring quality of life. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health.
Number of participants with malignant brain edema | 24 hour
  1) acute, complete MCA(middle cerebral artery) infarction with early parenchymal hypodensity of at least 50% of the MCA territory and signs of local brain swelling such as sulcal effacement and compression of the lateral ventricle; 2) midline shift of >5 mm at the septum pellucidum or pineal gland with obliteration of the basal cisterns; and 3) neurological deterioration consisting of a NIHSS increase by >2 points and decrease in the level of consciousness to a score of ≥ 1 on item 1A of the NIHSS.
Number of participants with treatment failure | 24 hour
  failure to achieve goal blood pressure(BP) for 2 consecutive BP measurements during the first 24 hours following EVT(endovascular thrombectomy)
CT or MRI ASPECTS(Alberta Stroke Program Early CT Score) | 36 hour
  Alberta Stroke Program Early CT Score(ASPECTS) is a 10-point quantitative score used to assess early ischemic changes on non-contrast CT head.
  To compute the ASPECTS, 1 point is subtracted from 10 for any evidence of early ischemic change for each of the defined regions. Identifying patients with a greater likelihood of poor functional outcome (scores <8) may be helpful in the early stages of care for supporting transfer or therapy decisions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Yonsei University College of Medicine, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
This is not a drug comparison study. Therefore IPD will not be shared.

REFERENCES:
- [Derived] Jung JW, Kim YD, Heo J, Lee H, Kim BM, Kim DJ, Shin NY, Joo H, Cho BH, Ahn SH, Park H, Sohn SI, Hong JH, Yun J, Song TJ, Chang Y, Kim GS, Seo KD, Lee K, Chang JY, Seo JH, Lee S, Baek JH, Cho HJ, Shin DH, Kim J, Yoo J, Baik M, Jung YH, Hwang YH, Kim CK, Kim JG, Lee IH, Choi JK, Lee CJ, Park S, Jeon S, Lee HS, Kim KH, Kwon SU, Bang OY, Heo JH, Nam HS; OPTIMAL-BP Trial Investigators. Association Between Intravenous Antihypertensives and Functional Outcome After Successful Endovascular Thrombectomy. Stroke. 2025 Sep;56(9):2503-2515. doi: 10.1161/STROKEAHA.125.051696. Epub 2025 Jul 3. PMID 40605757
- [Derived] Jung JW, Kim KH, Yun J, Joo H, Kim YD, Heo J, Lee H, Kim BM, Kim DJ, Shin NY, Cho BH, Ahn SH, Park H, Sohn SI, Hong JH, Song TJ, Chang Y, Kim GS, Seo KD, Lee K, Chang JY, Seo JH, Lee S, Baek JH, Cho HJ, Shin DH, Kim J, Yoo J, Baik M, Jung YH, Hwang YH, Kim CK, Kim JG, Lee IH, Choi JK, Lee CJ, Park S, Jeon S, Lee HS, Kwon SU, Bang OY, Heo JH, Nam HS. Blood pressure management based on infarct volume after successful endovascular thrombectomy. Eur Stroke J. 2025 Dec;10(4):1281-1291. doi: 10.1177/23969873251335204. Epub 2025 May 2. PMID 40317165
- [Derived] Yun J, Kim KH, Jung JW, Kim YD, Heo J, Lee H, Choi JK, Lim IH, Hong SH, Kim BM, Kim DJ, Shin NY, Cho BH, Ahn SH, Park H, Sohn SI, Hong JH, Song TJ, Chang Y, Kim GS, Seo KD, Lee K, Chang JY, Seo JH, Lee S, Baek JH, Cho HJ, Shin DH, Kim J, Yoo J, Baik M, Lee KY, Jung YH, Hwang YH, Kim CK, Kim JG, Lee CJ, Park S, Jeon S, Lee HS, Kwon SU, Lee IH, Bang OY, Heo JH, Nam HS. Effects of blood pressure lowering in patients treated with intravenous thrombolysis before endovascular thrombectomy. Int J Stroke. 2025 Jul;20(6):696-707. doi: 10.1177/17474930251315630. Epub 2025 Feb 6. PMID 39819210
- [Derived] Nam HS, Kim YD, Heo J, Lee H, Jung JW, Choi JK, Lee IH, Lim IH, Hong SH, Baik M, Kim BM, Kim DJ, Shin NY, Cho BH, Ahn SH, Park H, Sohn SI, Hong JH, Song TJ, Chang Y, Kim GS, Seo KD, Lee K, Chang JY, Seo JH, Lee S, Baek JH, Cho HJ, Shin DH, Kim J, Yoo J, Lee KY, Jung YH, Hwang YH, Kim CK, Kim JG, Lee CJ, Park S, Lee HS, Kwon SU, Bang OY, Anderson CS, Heo JH; OPTIMAL-BP Trial Investigators. Intensive vs Conventional Blood Pressure Lowering After Endovascular Thrombectomy in Acute Ischemic Stroke: The OPTIMAL-BP Randomized Clinical Trial. JAMA. 2023 Sep 5;330(9):832-842. doi: 10.1001/jama.2023.14590. PMID 37668619
- [Derived] Nam HS, Kim YD, Choi JK, Baik M, Kim BM, Kim DJ, Heo J, Shin DH, Lee KY, Jung YH, Baek JH, Hwang YH, Sohn SI, Hong JH, Park H, Kim CK, Kim GS, Seo KD, Lee K, Seo JH, Bang OY, Seo WK, Chung JW, Chang JY, Kwon SU, Lee J, Kim J, Yoo J, Song TJ, Ahn SH, Cho BH, Cho HJ, Kim JG, Chang Y, Lee CJ, Park S, Park G, Lee HS. Outcome in Patients Treated with Intra-arterial thrombectomy: The optiMAL Blood Pressure control (OPTIMAL-BP) Trial. Int J Stroke. 2022 Oct;17(8):931 - 937. doi: 10.1177/17474930211041213. Epub 2021 Aug 24. PMID 34427481
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37668619/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34427481/